CLINICAL TRIAL: NCT04215289
Title: Compatibility of Qnox Values With Hemodynamic Changes as a Predictor of Pain Response in Tracheal Intubation Procedures
Brief Title: Compatibility of Qnox Values With Hemodynamic Changes in Tracheal Intubation Procedures
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, MD, Indonesia University
Other Study IDs: IndonesiaUAnes 049
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Qnox Values as a Predictor of Pain Response
Keywords: qNox Values, Hemodynamic changes, Predictor of pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to analyze the compatibility of Qnox values with hemodynamic changes as a predictor of pain response in tracheal intubation procedures

DETAILED DESCRIPTION:
Fifty-four patients were given informed consent before enrolling the study. Non-invasive blood pressure monitor, electrocardiogram, pulse oxymetry, and Conox probe were set on the subjects in the operation room. Baseline hemodynamic is noted. General anesthesia induction was done by fentanyl 2.5 mcg/kg and propofol 2 mg/kg. Endotracheal tube intubation was facilitated with rocuronium 0.8 mg/kg as muscle relaxant. qNox values right before intubation and after intubation is noted, as well as hemodynamic changes in one minute after intubation

ELIGIBILITY:
Inclusion Criteria:

* patient undergoes general anesthesia with tracheal intubation
* fasting as required for surgery
* physical ASA status I - II
* signing informed consent

Exclusion Criteria:

* patient with difficult airway management
* patient with history of central nervous system abnormalities
* patient with history of hypersensitivity to drugs for general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients undergo general anesthesia procedure with tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Qnox Values | 1 minutes
  Observe the Qnox Values with Hemodynamic Changes to predict pain response

CONTACTS AND LOCATIONS:
Overall Officials: Adhrie Sugiarto, MD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griesdale DE, Bosma TL, Kurth T, Isac G, Chittock DR. Complications of endotracheal intubation in the critically ill. Intensive Care Med. 2008 Oct;34(10):1835-42. doi: 10.1007/s00134-008-1205-6. Epub 2008 Jul 5. PMID 18604519
- [Result] Ko DD, Kang H, Yang SY, Shin HY, Baek CW, Jung YH, Woo YC, Kim JY, Koo GH, Kim SD. A comparison of hemodynamic changes after endotracheal intubation by the Optiscope and the conventional laryngoscope. Korean J Anesthesiol. 2012 Aug;63(2):130-5. doi: 10.4097/kjae.2012.63.2.130. Epub 2012 Aug 14. PMID 22949980
- [Result] Jensen EW, Valencia JF, Lopez A, Anglada T, Agusti M, Ramos Y, Serra R, Jospin M, Pineda P, Gambus P. Monitoring hypnotic effect and nociception with two EEG-derived indices, qCON and qNOX, during general anaesthesia. Acta Anaesthesiol Scand. 2014 Sep;58(8):933-41. doi: 10.1111/aas.12359. Epub 2014 Jul 4. PMID 24995461
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Loeser JD, Treede RD. The Kyoto protocol of IASP Basic Pain Terminology. Pain. 2008 Jul 31;137(3):473-477. doi: 10.1016/j.pain.2008.04.025. Epub 2008 Jun 25. No abstract available. PMID 18583048